CLINICAL TRIAL: NCT07294287
Title: Impact of Microneedling on the Gingival Tissue Surrounding Implant Supported Fixed Restoration.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Al-Ahmady El-Meligy, Lecturer of Oral Medicine, Periodontology, Oral Diagnosis and Oral Radiology Faculty of Dentistry, Tanta University, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #R-FP-10-24-3150
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gingiva; Dental Implants
MeSH Terms: interventions — Angiopoietin-Like Protein 6

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel treatment groups:
  AGF alone. Microneedling combined with Accelerated Growth Factor (AGF) Each participant receives only one type of intervention, and the outcomes are compared between groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated Growth Factor (AGF) Injection Only (Active Comparator): Participants in this arm received autologous Accelerated Growth Factor (AGF) injection alone into the peri-implant mucosa (0.2-0.3 mL per site) in the maxillary anterior region, without prior microneedling. The AGF was prepared from 10 mL of venous blood via a standardized single-step centrifugation procedure to obtain a growth factor-rich fraction. Gingival thickness and soft tissue parameters were evaluated using the same intraoral scanner and transgingival file method at baseline, 3 months, and 6 months
  Interventions: Procedure: Accelerated Growth Factor (AGF) Injection Only
- Microneedling Combined with Accelerated Growth Factor (AGF) (Experimental): Participants in this arm received microneedling around the peri-implant mucosa in the maxillary anterior region using sterile disposable glucometer lancets under aseptic conditions. Repeated micro-perforations were created circumferentially until pinpoint bleeding appeared. Immediately afterward, autologous Accelerated Growth Factor (AGF) was injected (0.2-0.3 mL per site) into the treated mucosa. AGF was prepared from 10 mL of venous blood using a single-step centrifugation protocol to isolate the growth factor-rich fraction. Gingival thickness and soft tissue parameters were assessed using an intraoral scanner combined with a transgingival file measurement technique at baseline, 3 months, and 6 months.
  Interventions: Procedure: Microneedling Combined with Accelerated Growth Factor (AGF)

INTERVENTIONS:
Procedure: Microneedling Combined with Accelerated Growth Factor (AGF) — Participants in this arm received microneedling around the peri-implant mucosa in the maxillary anterior region using sterile disposable glucometer lancets under aseptic conditions. Repeated micro-perforations were created circumferentially until pinpoint bleeding appeared. Immediately afterward, autologous Accelerated Growth Factor (AGF) was injected (0.2-0.3 mL per site) into the treated mucosa. AGF was prepared from 10 mL of venous blood using a single-step centrifugation protocol to isolate the growth factor-rich fraction. Gingival thickness and soft tissue parameters were assessed using an intraoral scanner combined with a transgingival file measurement technique at baseline, 3 months, and 6 months.
  Arms: Microneedling Combined with Accelerated Growth Factor (AGF)
Procedure: Accelerated Growth Factor (AGF) Injection Only — Participants in this arm received autologous Accelerated Growth Factor (AGF) injection alone into the peri-implant mucosa (0.2-0.3 mL per site) in the maxillary anterior region, without prior microneedling. The AGF was prepared from 10 mL of venous blood via a standardized single-step centrifugation procedure to obtain a growth factor-rich fraction. Gingival thickness and soft tissue parameters were evaluated using the same intraoral scanner and transgingival file method at baseline, 3 months, and 6 months
  Arms: Accelerated Growth Factor (AGF) Injection Only

SUMMARY:
This randomized clinical trial aims to evaluate the effect of microneedling with and without accelerated growth factor (AGF) injection on gingival tissue surrounding implant-supported fixed restorations. The peri-implant soft tissue phenotype is an important determinant of long-term implant stability and esthetic success. Patients with thin gingival biotype are more susceptible to mucosal recession, soft tissue transparency, and peri-implant complications. Enhancing gingival thickness and keratinized tissue width using minimally invasive methods can improve esthetic and biological outcomes.

Microneedling has recently been proposed as a simple and minimally invasive approach that stimulates local healing by inducing controlled micro-injury. It triggers angiogenesis and the release of intrinsic growth factors that promote soft tissue regeneration. Accelerated Growth Factor (AGF) is an autologous platelet concentrate obtained through a single-step centrifugation technique. It contains a high concentration of platelet-derived and vascular growth factors that enhance tissue repair and collagen synthesis. Combining microneedling with AGF may therefore produce synergistic effects, improving the soft tissue phenotype and peri-implant mucosal stability.

The study will include 20 participants aged 18-34 years with thin gingival biotype (0.8-1 mm) around maxillary anterior implants. Participants will be randomly assigned to one of two groups:

1. AGF group: AGF injection alone.
2. Microneedling + AGF group: Microneedling using sterile disposable lancets until pinpoint bleeding occurs, followed by AGF injection (0.2-0.3 mL per site).

Clinical parameters including gingival thickness (GT), keratinized tissue width (KTW), probing depth (PD), and bleeding index (BI) will be recorded at baseline, 3 months, and 6 months. All participants will receive standardized zirconia restorations following osseointegration. Statistical analysis will include intra- and inter-group comparisons, with significance set at p < 0.05.

The study is expected to clarify whether combining microneedling with AGF enhances peri-implant soft tissue thickness more effectively than AGF alone. If successful, this combined minimally invasive approach may offer a practical and biologically based technique to improve soft tissue health and esthetics around dental implants.

DETAILED DESCRIPTION:
The peri-implant mucosa plays a crucial role in the biological and esthetic stability of dental implants. A thin gingival biotype is often associated with soft tissue recession, marginal bone loss, and esthetic compromise. Conventional augmentation techniques such as connective tissue grafting are effective but involve additional morbidity, donor site discomfort, and variable esthetic results. This study investigates a minimally invasive approach combining microneedling and accelerated growth factor (AGF) injection to enhance the gingival tissue phenotype around implant-supported restorations.

Microneedling is based on creating controlled micro-perforations in the soft tissue surface using fine needles. These micro-injuries induce a natural wound healing cascade that includes platelet activation, release of endogenous growth factors, angiogenesis, and fibroblast stimulation. The process enhances collagen deposition and epithelial thickening, which may increase the overall gingival thickness and keratinized tissue width.

AGF is an autologous blood-derived product obtained by a standardized single-step centrifugation technique that separates platelet-rich fractions containing high levels of biologically active molecules such as PDGF, VEGF, and TGF-β. These factors promote tissue regeneration and accelerate wound healing. Injecting AGF into peri-implant mucosa provides a reservoir of growth factors that stimulate fibroblast activity, improve tissue vascularity, and enhance collagen formation.

The hypothesis of this trial is that combining microneedling with AGF will yield superior soft tissue enhancement compared to AGF alone.

Study Design

This is a prospective, randomized, single-blinded, parallel-arm interventional clinical trial. 20 sites for patients aged 18-34 years with thin gingival biotype (0.8-1mm) in the maxillary anterior region will be included. Participants will be randomly assigned to two groups using a computer-generated random sequence:

1. AGF Group: AGF injection only.
2. Microneedling + AGF Group: Microneedling using sterile disposable lancets until pinpoint bleeding occurs, immediately followed by AGF injection (0.2-0.3 mL per site).

Methodology

The study follows five sequential phases:

1. Pre-surgical Phase: Clinical and radiographic evaluation, oral hygiene instructions, baseline measurement of GT, KTW, PD, and BI.
2. Surgical Phase: Implant placement in the maxillary anterior region followed by 3-4 months of osseointegration.
3. Intervention Phase: Randomized treatment application after healing.
4. Restorative Phase: Fabrication and cementation of standardized zirconia crowns.
5. Follow-up Phase: Assessment of all parameters at baseline, 3, and 6 months. Outcome Measures

   * Primary Outcome: Gingival thickness (GT) at baseline, 3, and 6 months.
   * Secondary Outcomes: Keratinized tissue width (KTW), probing depth (PD), and bleeding index (BI).

Statistical Analysis Data will be analyzed using SPSS software (IBM). Paired and unpaired t-tests will compare intra- and inter-group differences. The significance level will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-34 years
* Thin gingival biotype ( 0.8- 1mm GT at maxillary anterior teeth)
* Non-smokers
* Plaque index (PI) score 0-1
* No bleeding on probing
* No malocclusion or crowding affecting implant site

Exclusion Criteria:

* Active orthodontic treatment
* Previous periodontal surgery at study sites
* Systemic diseases affecting healing
* Use of anticoagulants or drugs causing gingival enlargement
* Mucogingival stress or bruxism

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-05 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Gingival thickness (GT) | Baseline, 3 months, and 6 months after intervention
  Gingival thickness will be measured to assess the effect of accelerated growth factor injection with and without microneedling on peri-implant soft tissue phenotype.
  Measurements will be taken at the mid-facial point of the implant site using a transgingival file technique combined with digital evaluation via intraoral scanning to ensure accuracy and reproducibility.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa M Elgendy, lecturer, Study Chair — Lecturer of prosthodontics, faculty of dentistry, Tanta university, Egypt.; Shimaa M Eltantawy, lecturer, Principal Investigator — Lecturer of fixed prosthodontics, Faculty of Dentistry, Tanta University, Egypt; Ahmed A Mosleh, lecturer, Study Director — Lecturer of oral and maxillofacial surgery, Faculty of Dentistry, Tanta University, Egypt
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toita T. [Uterine cervical cancer]. Nihon Igaku Hoshasen Gakkai Zasshi. 2002 Apr;62(5):198-201. Japanese. PMID 12043223
- [Background] Ozsagir ZB, Saglam E, Sen Yilmaz B, Choukroun J, Tunali M. Injectable platelet-rich fibrin and microneedling for gingival augmentation in thin periodontal phenotype: A randomized controlled clinical trial. J Clin Periodontol. 2020 Apr;47(4):489-499. doi: 10.1111/jcpe.13247. Epub 2020 Feb 11. PMID 31912532